CLINICAL TRIAL: NCT06881446
Title: Immune Checkpoint Inhibitors and Anti-vascular Endothelial Growth Factor Antibody/tyrosine Kinase Inhibitors with or Without Transarterial Chemoembolization As First-line Treatment for Advanced Hepatocellular Carcinoma with Vascular Invasions
Brief Title: Immune Checkpoint Inhibitors and Anti-vascular Endothelial Growth Factor Antibody/tyrosine Kinase Inhibitors with or Without TACE for Advanced HCC with Vascular Invasions
Status: Recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Other Study IDs: CHANCE2505
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: transarterial chemoembolization; hepatocellular carcinoma; immune checkpoint inhibitors; molecular target therapies
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Immune checkpoint inhibitors and anti-vascular endothelial growth factor antibody/tyrosine kinase inhibitors with or without transarterial chemoembolization as first-line treatment for advanced hepatocellular carcinoma with vascular invasions

DETAILED DESCRIPTION:
The vascular invasions is a common complication in 16% to 30% of patients with hepatocellular carcinoma (HCC), contributing to poor prognosis and increasing the risk of cancer recurrence, with a median survival of approximately 2.7 to 4 months without intervention. Both the European Association for the Study of the Liver and the American Association for the Study of Liver Diseases guidelines recommend that HCC patients with vascular invasions be classified as Barcelona Clinic Liver Cancer Stage C and receive systemic treatments. Nevertheless, there is limited data on patients with highly complicated HCC and no optimal treatment strategy for this patient population. Tyrosine kinase inhibitors (TKIs) and immune checkpoint inhibitors (ICIs) are commonly utilized in the systemic therapy of HCC, while the combination of transcatheter arterial chemoembolization (TACE) with systemic therapy has significantly improved treatment outcomes in advanced-stage patients. Therefore, we hypothesized that a triplet regimen comprising TACE, TKI, and ICIs may yield better prognoses for HCC patients with vascular invasions. This study aims to compare the safety and efficacy of the triplet regimen of TKIs, ICIs, and TACE versus Lenvatinib combined with ICIs in advanced-stage HCC with vascular invasions

ELIGIBILITY:
1. Has a diagnosis of HCC confirmed by radiology, histology, or cytology;
2. Barcelona Clinic Liver Cancer (BCLC) stage C with the presence of macrovascular invasion;
3. Has not received any previous systemic therapy for HCC (including chemotherapy, molecularly targeted therapy, immunotherapy);
4. Both PD-1/PD-L1 inhibitors and anti-angiogenesis drugs patients received only include marketed drugs but are not limited to HCC approval;
5. TACE was performed after the first PD-1/PD-L1 inhibitor/anti-angiogenic drug treatment or before treatment (within 3 months);
6. Received at least 1 cycle of PD-1/PD-L1 inhibitor/anti-angiogenic drug combination therapy after TACE treatment;
7. Has repeated measurable intrahepatic lesions;

Exclusion Criteria:

1. Cholangiocarcinoma, fibrolamellar, sarcomatoid hepatocellular carcinoma, and mixed hepatocellular/cholangiocarcinoma subtypes(confirmed by histology, or pathology) are not eligible;
2. Unable to meet criteria of combination timeframe described above;
3. Child-Pugh C or PS>2 or Severe hepatic encephalopathy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with advanced HCC who received TACE in combination with PD-1/PD-L1 inhibitors and molecular target therapies under real-world practice conditions
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | up to approximately 2 years
  The OS is defined as the time from the initiation of any combination treatment to death due to any cause.
Progression free survival(PFS) according to per mRECIST or RECIST 1.1 | up to approximately 2 years
  per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Description: The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to RECIST 1.1) or death due to any cause, whichever occurs first.
  PFS per Modified Response Evaluation Criteria in Solid Tumors (mRECIST) Description: The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to mRECIST) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
ORR per mRECIST | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented CR or PR per mRECIST
Objective response rate(ORR) per RESCIST 1.1 | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per RECIST 1.1.
Adverse event(AE) per Common Terminology Criteria for Adverse Events(CTCAE) 5.0 | up to approximately 2 years
  The percentage and degree of patients who experience at least one AE, whether or not considered related to the treatment, according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, M.D, Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China